CLINICAL TRIAL: NCT06490861
Title: An Open Multi-centre Investigation to Evaluate the Performance of the Paragit Sleeve With build-in sEMG Sensors, Kinetic Sensors, and Smart-textile to Measure and Monitor Motor Symptoms and Treatment-induced Dyskinesia in Patients With Parkinson's Disease
Brief Title: Performance of the Paragit Sleeve to Measure and Monitor Motor Symptoms in Patients With Parkinson's Disease
Acronym: PARPIV23
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Paragit ApS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PARPIV23
Record Dates: First submitted 2024-06-13; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paragit (Experimental): Sleeve to quantify symptoms
  Interventions: Device: Paragit

INTERVENTIONS:
Device: Paragit — Sleeve to quantify symptoms

SUMMARY:
This investigation is undertaken to:

* Evaluate the accuracy and reliability of the device in measuring and recording motor symptoms associated with Parkinson's Disease (PD), and
* To assess the safety and tolerability of the device in patients with PD.

ELIGIBILITY:
Inclusion Criteria:

1. Parkinson disease: Clinically diagnosed
2. Age ≥ 50 (not in the childbearing aged as defined by Statistics Denmark, 15-49)
3. Experiencing at least two of following symptoms and/or side effect on a daily basis:

   * Rigidity
   * Tremor
   * Bradykinesia
   * Dyskinesia (treatment side effect)
4. Provision of informed consent, i.e., the subject must be able to:

   * Read and understand the Patient Information and Consent Form
   * Sign the Patient Information and Consent Form.

Exclusion Criteria:

1. Known allergy/hypersensitivity to any material in direct contact with the skin (stainless steel, silicone and polyester)
2. MMSE <24
3. Other neurological diseases

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Tremor | During the clinical assessment, and for the following 24h.
  Tremor will be assessed using the device, measured with superficial EMG [Volts], and inertial measurement unit [m/s2]. Correlation with clinical gold-standard (MDS-UPDRS) will be studied.
Bradykinesia | During the clinical assessment, and for the following 24h.
  Bradykinesia will be assessed using the device, measured inertial measurement unit [m/s2]. Correlation with clinical gold-standard (MDS-UPDRS) will be studied.
Rigidity | During the clinical assessment, and for the following 24h.
  The device will assess rigidity, measured with superficial EMG [Volts], and inertial measurement unit [m/s2]. Correlation with clinical gold-standard (MDS-UPDRS) will be studied.
Dyskinesia | During the clinical assessment, and for the following 24h.
  The device will assess rigidity, measured with superficial EMG [Volts], and inertial measurement unit [m/s2]. Correlation with clinical gold-standard (MDS-UPDRS) will be studied.

SECONDARY OUTCOMES:
Safety | During the clinical assessment , and for the following 24h.
  Safety of the Paragit Sleeve by assessment of device deficiencies and adverse events, non-serious and serious, rated for causality.
Usability | During the clinical assessment , and for the following 24h.
  The usability of the device will be studied using a questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Beata María Ana, Madrid, Spain